CLINICAL TRIAL: NCT06343935
Title: A National Multicenter, Real-world Study of Linperlisib in the Treatment of Lymphoma
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YY-20394-014
Record Dates: First submitted 2024-03-25; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Indolent B-cell Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group(linperlisib 80mg qd) (Experimental): After enrollment, the patients in treatment group were orally administered with a starting dose of 80mg qd for 21 days. On the 21st day of the 4th cycle, if the patient has no tumor progression and no intolerable toxicity, after the researcher determines that the drug therapy can be continued, the patient should take linperlisib 80mg qd for two consecutive weeks per cycle and stop taking it for one week, and conduct regular safety and tumor efficacy evaluation until the disease progresses, toxicity becomes intolerable or the researcher determines that it is not suitable to continue treatment. The maximum duration of treatment is two years.
  Interventions: Drug: Linperlisib
- control group(linperlisib 80mg 14d-on 7d-off) (Experimental): In the control group, patients were orally administered at the starting dose of 80mg qd for 21 days after enrollment. On the 21st day of the 4th cycle, if the patient has no tumor progression and no intolerable toxicity, the patient will continue to receive Linperlisib 80mg qd after the investigator determines that the drug therapy can be continued, and the safety and tumor efficacy evaluation will be conducted regularly until the disease progresses, toxicity becomes intolerable, or the investigator determines that the treatment is not suitable for further treatment. The maximum duration of treatment is two years.
  Interventions: Drug: Linperlisib

INTERVENTIONS:
Drug: Linperlisib — Linperlisib is a small molecule inhibitor of phosphoinositol 3-kinase-δ (PI3K-δ)
  Other Names: YY-20394

SUMMARY:
This is a national multicenter, randomized controlled, open, dose-optimized Phase IV study. It is expected to enroll approximately 88 patients with relapsed/refractory indolent B-cell lymphoma. The aim is to evaluate the efficacy and safety of linperlisib in the treatment of patients with relapsed/refractory indolent B-cell lymphoma at two doses/modes of administration (clinically recommended dose/mode and optimized dose/mode).

DETAILED DESCRIPTION:
This is a national multicenter, randomized controlled, open, dose-optimized Phase IV study. It is expected to enroll approximately 88 patients with relapsed/refractory indolent B-cell lymphoma. The aim is to evaluate the efficacy and safety of linperlisib in the treatment of patients with relapsed/refractory indolent B-cell lymphoma at two doses/modes of administration (clinically recommended dose/mode and optimized dose/mode).

Patients were divided to two groups by stratified randomization according to tumor type (FL, CLL/SLL, MZL, others) during the screening period. Both groups were orally administered with a starting dose of 80mg qd for 21 days. On the 21st day of the 4th cycle, if the patient's tumor does not progress and there is no intolerable toxicity, after the researchers determined that medication could be continued, one group of patients continued to take 80mg qd dose continuously, and the other group of patients continued to take 80mg qd dose continuously for two weeks per cycle and stopped for one week, and safety and tumor efficacy evaluation were conducted regularly. The maximum duration of treatment is two years until the disease progresses, toxicity becomes intolerable, or the investigator determines that it is not appropriate to continue treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with r/r indolent B-cell lymphoma confirmed by histology or cytology, mainly follicular lymphoma (FL), chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), marginal zone B-cell lymphoma (MZL), and lymphoplasmacytic lymphoma/macroglobulinemia (LPL/WM),
2. ECOG performance status (PS) 0 ~ 2 points,
3. Expected survival ≥3 months,

5) At least one measurable lesion was present in patients other than CLL, LPL/WM; 6) Good organ function level, 7) The elution period from the end of previous anti-tumor therapy (including radiotherapy, chemotherapy, immunotherapy, surgery or molecular targeted therapy) to participation in this trial is ≥4 weeks, in which the elution period of small-molecule targeted drugs and Chinese medicines with anti-tumor effects is ≥14 days.

Exclusion Criteria:

1. Those who have progressed with antitumor drugs targeting PI3Kδ (except for those who cannot tolerate them),
2. There is a third space effusion (such as a large amount of pleural fluid and ascites) that the investigators judge to be uncontrollable,
3. Steroid hormone dosage (equivalent amount of prednisone) was greater than 20mg/ day for 4 weeks before enrollment, and continuous use was more than 14 days,
4. Inability to swallow, chronic diarrhea or intestinal obstruction, there are multiple factors that affect drug use and absorption,
5. Allergic constitution, or known allergic history of the drug components,
6. Patients with active viral, bacterial or fungal infections (such as pneumonia) within 4 weeks prior to enrollment; Or had uncontrolled pulmonary fibrosis, acute lung disease, or interstitial lung disease within 4 weeks prior to enrollment,
7. Infected with HBV and HCV,
8. History of immune deficiency,
9. Moderate or severe heart disease,
10. Have undergone major surgery within 28 days before signing informed consent, or plan to undergo major surgery during the study period,
11. The first study of patients with a history of other malignancies within 5 years prior to drug administration (except for patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, cervical carcinoma in situ, or other cancers in situ without disease recurrence within 2 years),
12. Received autologous hematopoietic stem cell transplantation within 90 days before the first medication,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From the first dose to the date of disease progression or date of death from any cause, whichever comes first，up to 24months
  The time from the first dose of study treatment to first documented disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective response rate | From the first dose to the date of disease progression or date of death from any cause, whichever comes first，up to 24months
  The proportion of subjects who have a Complete Response or Partial Response
Overall survival | From the first dose to the date of death from any cause, whichever comes first，up to 24months
  The time from the first dose of study treatment to death for any reason.
Adverse event | From enrollment receiving Linperlisib to 30 days after the last linperlisib treatment.
  Incidence of adverse events evaluated by NCI CTCAE v5.0 and associated dose of linperlisib
Serious adverse event | From enrollment receiving Linperlisib to 30 days after the last linperlisib treatment.
  Incidence of serious adverse event and associated dose of linperlisib

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, Principal Investigator — Hematology Tumor Research Center of Harbin First Hospital